CLINICAL TRIAL: NCT00909012
Title: Quantitative Requirements of Docosahexaenoic Acid for Neural Function in Children With Phenylketonuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Prof. Berthold Koletzko, Prof., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 455-08
Record Dates: First submitted 2009-04-22; First posted 2009-05-27 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Phenylketonuria
Keywords: phenylketonuria; docosahexaenoic acid; visually evoked potential; choice-reaction time
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: high oleic sunflower oil
- 2 (Experimental)
  Interventions: Dietary Supplement: microalgal oil
- 3 (Experimental)
  Interventions: Dietary Supplement: microalgal oil
- 4 (Experimental)
  Interventions: Dietary Supplement: microalgal oil
- 5 (Experimental)
  Interventions: Dietary Supplement: microalgal oil

INTERVENTIONS:
Dietary Supplement: high oleic sunflower oil — placebo, which does not provide DHA
  Arms: 1
Dietary Supplement: microalgal oil — the supplement provides 20 mg DHA per capsule (1 or 2 are consumed per day, depending on body weight)
  Arms: 2
Dietary Supplement: microalgal oil — the supplement provides 40 mg DHA per capsule (1 or 2 are consumed per day, depending on body weight)
  Arms: 3
Dietary Supplement: microalgal oil — the supplement provides 80 mg DHA per capsule (1 or 2 are consumed per day, depending on body weight)
  Arms: 4
Dietary Supplement: microalgal oil — the supplement provides 130 mg DHA per capsule (1 or 2 are consumed per day, depending on body weight)
  Arms: 5

SUMMARY:
Patients with phenylketonuria (PKU) have an inborn error in the metabolism of the amino acid phenylalanine (Phe) and thus must follow a strictly controlled protein-restricted diet from early infancy. This protein-restricted diet is devoid of natural dietary sources of n-3 long chain polyunsaturated fatty acids (LC-PUFA), such as eggs, meat, milk or fish. Therefore, blood concentrations of n-3 LC-PUFA, especially of docosahexaenoic acid (DHA) are reduced in PKU children compared to healthy controls. DHA availability is considered important for optimal neurological function. Previous studies have shown that neural function of PKU children is improved by high dose supplementation of fish oil providing DHA, as shown by significant improvements of both visual evoked potential latencies and of fine motor skills and coordination, but no dose response relationship has been established so far.

This multicentric double-blind randomized trial aims at determining quantitative DHA requirements for optimal neural function in PKU children. Patients with classical PKU from several major treatment centers in Europe will be randomized to receive between 0 and 8 mg of DHA per kg body weight daily for a duration of 6 months. Biochemical (fatty acid composition of plasma phospholipids, lipoprotein metabolism and metabolic profiles), and functional testing (visual evoked potentials, fine motor skills, cognitive function and markers of immune function) will be performed at baseline and after 6 months. Intake per kg body weight will be related to outcome parameters and thus a possible dose response relationship will be defined. The results from this study are expected to contribute to the improvement of the diet of PKU patients, but they also have the potential to help defining quantitative DHA needs of healthy children.

The primary hypothesis is that supplementation with DHA improves visual function in children with PKU.

ELIGIBILITY:
Inclusion Criteria:

* Children with classical PKU, who have been diagnosed and treated from the newborn period onwards
* Classical PKU must have been established by a baseline plasma phenylalanine (PHE) level >1200 µmol/L or detection of underlying mutations
* Children are clinically healthy besides classical PKU
* Good metabolic control (a minimum of 2 Phe-values during the last 6 months are needed with average Phe values being below 480 µmol/L in the last 6 months)
* No n-3 LC-PUFA supplementation for at least 6 months before enrolment
* Written informed consent of parents exists

Exclusion Criteria:

* Severe neurological symptoms
* History of neurological disease
* Children are unable to take DHA-capsules regularly
* Acute illness, especially infections at the time of clinical examination/testing
* Children with weight/height over the 97th percentile or below the 3rd percentile
* Known hypersensitivity to fish oil products

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
latency of visually evoked potentials | assessed basally (before intervention start) and at the end of the 6 month intervention period

SECONDARY OUTCOMES:
fatty acid composition of plasma phospholipids | assessed basally (before intervention start) and at the end of the 6 month intervention period
fine motor skills | assessed basally (before intervention start) and at the end of the 6 month intervention period
test of reaction time | assessed basally (before intervention start) and at the end of the 6 month intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Principal Investigator — Dr. von Hauner Children Hospital, Ludwig-Maximilians-Universitaet Muenchen
Locations (6):
- Germany (2):
  - Zentrum für Kinder- und Jugendmedizin, Heidelberg
  - LMU, München
- Department of Pediatrics, San Paolo Hospital Milano, Milan, Italy
- Department of Pediatrics, IFIMAV-Hospital M. Valdecill, Santander, Spain
- United Kingdom (2):
  - The Childrens Hospital Birmingham, Birmingham
  - Department of Pediatrics, Great Ormond Street Hospital for Sick Children, London

REFERENCES:
- [Result] Demmelmair H, MacDonald A, Kotzaeridou U, Burgard P, Gonzalez-Lamuno D, Verduci E, Ersoy M, Gokcay G, Alyanak B, Reischl E, Muller-Felber W, Faber FL, Handel U, Paci S, Koletzko B. Determinants of Plasma Docosahexaenoic Acid Levels and Their Relationship to Neurological and Cognitive Functions in PKU Patients: A Double Blind Randomized Supplementation Study. Nutrients. 2018 Dec 7;10(12):1944. doi: 10.3390/nu10121944. PMID 30544518